CLINICAL TRIAL: NCT01846013
Title: Increasing Workplace Physical Activity in Sedentary Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1212M25961; UL1TR000114 (NIH)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Sit-Stand Workstations
Keywords: Sit-Stand Workstations; Increase Workplace Physical Activity
MeSH Terms: interventions — Stil protein, Drosophila

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stand (Experimental)
  Interventions: Behavioral: Stand
- Move (Experimental)
  Interventions: Behavioral: Move
- Stand and Move (Experimental)
  Interventions: Behavioral: Stand and Move
- General Wellness (No Intervention)

INTERVENTIONS:
Behavioral: Stand — Stand at least half of the workday at work.
  Arms: Stand
Behavioral: Move — Increase movement time at work. Move more by making small changes (walking meetings, take stairs, etc).
  Arms: Move
Behavioral: Stand and Move — Increase standing time to half of workday (4h) and increase movement time at work.
  Arms: Stand and Move

SUMMARY:
Purpose:

The purpose of this study is to implement and evaluate a randomized controlled trial in sitting office workers to reduce sitting time through the use of motorized and non-motorized sit/stand workstations as well as a walking intervention.

Hypotheses:

1. Compared to the control group, total physical activity will be higher in the standing and walking intervention groups.
2. The combined standing and walking group will have higher total physical activity than the other three groups.
3. Compared to the control group, the fitness and health outcomes will be improved for the standing and walking groups.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary adults who use a single computer workstation for the majority of their workday
* Work full time (at least 35 hours per week)
* Must have ability to safely begin a standing and/or walking protocol with no adverse side effects

Exclusion Criteria:

* Musculoskeletal or joint problems
* Severe autoimmune conditions
* Varicose veins that may cause pain
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Total physical activity | 6-months

SECONDARY OUTCOMES:
Fasting blood glucose | 6-months

OTHER OUTCOMES:
Total cholesterol | 6-months
Body composition | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Pereira, PhD, Principal Investigator — University of Minnesota; Katie C Carpenter, PhD, Principal Investigator — University of Minnesota; Amanda R Bonikowske, MA, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - Fairview Energy Park, Saint Paul, Minnesota
  - MN Department of Human Services, Saint Paul, Minnesota